CLINICAL TRIAL: NCT01528111
Title: A Phase 1/2a, Randomized, Parallel-group, Double-masked, Vehicle-controlled, Dose-frequency Escalation Study to Evaluate the Safety, Tolerability, and Intraocular Pressure (IOP)-Lowering Efficacy of Topically Administered LX7101 in Subjects Diagnosed With Primary Open-angle Glaucoma (POAG) or Ocular Hypertension (OHT)
Brief Title: Study to Evaluate the Safety, Tolerability, and Efficacy of LX7101 in Subjects With Primary Open-angle Glaucoma or Ocular Hypertension
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Lexicon Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LX7101.7-101-OAG; LX7101.101 (Other: Lexicon Pharmaceuticals, Inc.)
Record Dates: First submitted 2012-02-03; First posted 2012-02-07 (Estimated); Last update posted 2015-09-14 (Estimated); Status verified 2015-08

CONDITIONS: Primary Open-angle Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — LX-7101

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Low dose LX7101 (Experimental): Days 1-3: once daily dose in study eye (eye with highest IOP); Days 4-7: once daily dose in study eye (eye with highest IOP) and fellow eye (other eye); Days 8-14: twice daily dose in study eye (eye with highest IOP) and fellow eye (other eye)
  Interventions: Drug: LX7101 (0.125%)
- High dose LX7101 (Experimental): Days 1-3: once daily dose in study eye (eye with highest IOP); Days 4-7: once daily dose in study eye (eye with highest IOP) and fellow eye (other eye); Days 8-14: twice daily dose in study eye (eye with highest IOP) and fellow eye (other eye)
  Interventions: Drug: LX7101 (0.25%)
- LX7101 Vehicle (Placebo Comparator): Days 1-3: once daily dose in study eye (eye with highest IOP); Days 4-7: once daily dose in study eye (eye with highest IOP) and fellow eye (other eye); Days 8-14: twice daily dose in study eye (eye with highest IOP) and fellow eye (other eye)
  Interventions: Drug: LX7101 Vehicle

INTERVENTIONS:
Drug: LX7101 (0.125%) — Subjects will receive 0.125% LX7101
  Arms: Low dose LX7101
Drug: LX7101 (0.25%) — Subjects will receive 0.25% LX7101
  Arms: High dose LX7101
Drug: LX7101 Vehicle — Subjects will receive vehicle
  Arms: LX7101 Vehicle

SUMMARY:
This Phase 1/2a study is intended to assess the safety, tolerability, and effects on intraocular pressure of two dose levels and two dose frequencies of LX7101 when administered topically in the eyes of patients diagnosed with primary open-angle glaucoma or ocular hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years of age
* Documented diagnosis of POAG or OHT, in both eyes
* Willing and able to provide written informed consent

Exclusion Criteria:

* History of any form of glaucoma in either eye, other than POAG
* Subjects who are unwilling or unable to discontinue contact lens wear prior to and during study
* History of ocular trauma in either eye <6 months prior to Screening
* History of ocular infection or ocular inflammation in either eye <3 months prior to Screening
* History of chronic or recurrent severe inflammatory eye disease, any severe ocular pathology, or clinically relevant or progressive retinal diseases in either eye
* Clinically relevant, severe central visual field loss, or documented significant progression of a visual field defect within 6 months prior to Screening in either eye
* Use of any ocular hypertensive medications (if applicable), in either eye, during the washout period and for the duration of the study
* Use of any glucocorticoid medications <2 weeks prior to Screening and throughout the duration of the study
* Use of any medication or substance on a chronic basis which has not been taken at a stable dose for at least 30 days prior to Screening
* Use of any nondiagnostic, topical, ophthalmic preparations, in either eye, other than artificial tears
* The presence of any concurrent condition or clinically significant laboratory findings at Screening that may interfere with any aspect of safety, study conduct, or interpretation of results
* Women who are pregnant or breast feeding
* Inability or difficulty instilling eye drops

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2012-03; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Number of subjects experiencing an adverse event | 15 Days

SECONDARY OUTCOMES:
Mean Intraocular Pressure (IOP) in the study eye | Days 1, 3, 7, 10, 14, 15
Best Corrected Visual Acuity (BCVA) | Days 1, 3, 7, 10, 14, 15
Slit lamp biomicroscopy exam (SLE) | Days 1, 3, 7, 10, 14, 15

CONTACTS AND LOCATIONS:
Overall Officials: Joel Freiman, M.D., MPH, Study Director — Lexicon Pharmaceuticals, Inc.
Locations (5):
- United States (5):
  - Lexicon Investigational Site, Morrow, Georgia
  - Lexicon Investigational Site, Memphis, Tennessee
  - Lexicon Investigational Site, Austin, Texas
  - Lexicon Investigational Site, Houston, Texas
  - Lexicon Investigational Site, San Antonio, Texas